CLINICAL TRIAL: NCT07386470
Title: Effect of Costoclavicular Versus Lateral Sagittal Infraclavicular Block on Hemidiaphragmatic Function: A Randomized Clinical Study
Brief Title: Comparison of Costoclavicular and Lateral Sagittal Infraclavicular Blocks
Acronym: CCLS-ICB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İrfan GUNGOR, MD, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICB-CC-LS-2022
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hemidiaphragmatic Paralysis; Upper Extremity Surgery
Keywords: Infraclavicular brachial plexus block; hemidiaphragmatic paralysis; costoclavicular brachial plexus block

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized, parallel group study comparing two ultrasound guided infraclavicular block techniques
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costoclavicular infraclavicular block (Experimental): Ultrasound-guided costoclavicular infraclavicular brachial plexus block
  Interventions: Procedure: Ultrasound-guided Infraclavicular block
- Lateral sagittal infraclavicular block (Active Comparator): Ultrasound-guided lateral sagittal infraclavicular brachial plexus block
  Interventions: Procedure: Ultrasound-guided Infraclavicular block

INTERVENTIONS:
Procedure: Ultrasound-guided Infraclavicular block — Ultrasound-guided infraclavicular brachial plexus block performed using either the costoclavicular or lateral sagittal approach with standardized local anesthetic volume.
  Other Names: costoclavicular infraclavicular block; lateral sagital infraclavicular block

SUMMARY:
This randomized clinical study aims to compare the effects of two different ultrasound-guided infraclavicular brachial plexus block techniques-costoclavicular and lateral sagittal approaches-in patients undergoing forearm, wrist, or hand surgery.

The primary objective of the study is to evaluate and compare the incidence of hemidiaphragmatic dysfunction associated with these two block techniques. Secondary outcomes include sensory and motor block characteristics, postoperative pain scores, analgesic requirements, and potential block-related complications.

Eligible adult patients scheduled for elective forearm or hand surgery are randomly assigned to receive either a costoclavicular or a lateral sagittal infraclavicular nerve block using bupivacaine under ultrasound guidance. Standard general anesthesia and postoperative analgesia protocols are applied.

The results of this study are expected to provide evidence on the relative safety and efficacy of these two infraclavicular block approaches, particularly regarding diaphragmatic function, and to help guide anesthesiologists in selecting the most appropriate regional anesthesia technique for upper extremity surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years
* ASA physical status I-III
* Scheduled for forearm, wrist, or hand surgery
* Planned infraclavicular brachial plexus block

Exclusion Criteria:

* Refusal of regional anesthesia
* Known allergy to local anesthetics
* Infection at the block site
* Pre-existing neurological deficit in the operative limb
* Severe pulmonary disease
* Coagulopathy or sepsis
* BMI > 40 kg/m²
* Psychiatric disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic excursion | Baseline(pre-block) and 30 minutes after block performance.
  Diaphragmatic excursion measured by ultrasound during normal and deep breathing to asses the effect of costoclavicular and lateral sagittal infraclavicular block techniques.

SECONDARY OUTCOMES:
Sensory and motor block onset time | Within the first 30 minutes after block performance.
  Time from completion of the infraclavicular block to achievement of complete sensory and motor block in the radial, median, ulnar, and musculocutaneous nerve distributions. Sensory and motor function were assessed every 5 minutes for up to 30 minutes after block performance, and block onset time was defined as the time to complete block.
Time to first postoperative analgesic requirement | Within the first 24 hours postoperatively.
  Time from the end of the surgery to the first analgesic requirement.

CONTACTS AND LOCATIONS:
Overall Officials: Irfan Güngör, MD, Principal Investigator — Gazi University Faculty of Medicine
Locations (1):
- Gazi University Faculty of Medicine, Department of Anesthesiology and Reanimation, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No